CLINICAL TRIAL: NCT01121991
Title: A Phase III, Multicentre, Open-label Prospective Study to Evaluate the Addition of Subcutaneous Recombinant Human-Luteinizing Hormone (Luveris) With r-hFSH on Follicular Development in Women Undergoing Ovarian Stimulation for ART
Brief Title: A Prospective Study to Evaluate the Addition of Subcutaneous Recombinant Human-Luteinizing Hormone With Recombinant Human-Follicle Stimulating Hormone on Follicular Development in Women Undergoing Ovarian Stimulation for Assisted Reproductive Technologies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Irene Kavanagh, Medical Research Manager, EMD Serono Canada Inc., an affiliate of Merck KGaA, Darmstadt, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMP 25244
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2011-03-18 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Infertility; Ovarian Stimulation
Keywords: Infertility; Ovarian Stimulation; Luveris; Lutropin alpha; Controlled ovarian stimulation; Reproductive techniques, assisted
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — Luteinizing Hormone, beta Subunit

INTERVENTIONS:
Drug: Recombinant Human-Luteinizing Hormone (Luveris) — Recombinant Human-Luteinizing Hormone (Luveris) was administered once daily subcutaneously at a starting dose of 150 IU per day beginning on stimulation Day 6.

SUMMARY:
In-vitro fertilization (IVF) of human oocytes followed by the replacement of embryo in the uterine cavity has become a well established treatment for female infertility attributable to damaged fallopian tubes, endometriosis or unexplained causes where alternative forms of therapy have failed. The most commonly used protocols of follicular stimulation now employs follicle stimulating hormone (FSH) and long-acting agonists of gonadotropin releasing hormone (GnRH) to prevent the occurrence of a mid-cycle luteinizing hormone (LH) surge and to ensure the induction of well-synchronized larger cohort of ovarian follicles.

The results of a number of studies have demonstrated that in the majority of clinical situations, FSH administration alone is sufficient to achieve successful follicular development. A study had shown that in subjects receiving recombinant human-follicle stimulating hormone (r-hFSH) and recombinant human-luteinizing hormone (r-hLH), pregnancy rates were similar in the younger and older age groups, however, in women receiving r-hFSH alone, there was a significant decline in pregnancy rates for women 35 and older. This particular study also went on to show that the subgroup of women 35 and older, may benefit from supplementary r-hLH. A number of studies have been conducted to assess the safety and efficacy of r-hLH administered concomitantly with r-hFSH in the presence of developing follicles to reduce the rate of growth of intermediate and small follicles while allowing the dominant follicle to continue to progress.

This was a Phase III, open-label, multicentre study to evaluate safety and efficacy of addition of Recombinant Human-Luteinizing Hormone (Luveris) to a standard assisted reproductive technologies (ART) protocol.

DETAILED DESCRIPTION:
Luteinizing hormone is a heterodimeric glycoprotein composed of a non-covalent association of an α and a β subunit. Prior to the generation of human-LH (hLH) through recombinant technology, hLH had only been available for therapeutic use as human menopausal gonadotropins (hMG), a co-extracted, purified preparation of hLH and hFSH from urine of post menopausal women. Recombinant Human-Luteinizing Hormone (Luveris) has been found to be well tolerated in human pharmacokinetic and pharmacodynamic studies at doses of up to 40,000 IU in healthy female volunteers without any Serious Adverse Event (SAE) experience being reported.

OBJECTIVES

* To evaluate safety and efficacy of addition of Recombinant Human-Luteinizing Hormone (Luveris) to a standard ART procedure.

In this study, subjects were first treated with a GnRH agonist to induce pituitary desensitization according to centre's standard practice followed by administration of r-hFSH. All subjects were then treated with Recombinant Human -Luteinizing Hormone (Luveris)150 IU per day subcutaneous (s.c.) from Day 6 of stimulation of their ART treatment cycle, continuing at the same dose until injection of hCG upto and including day of last FSH dose.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects who underwent ovarian stimulation for ART (IVF/ICSI) using r-hFSH.
* Subjects who in the opinion of the treating investigator met any of the following criteria to require r-LH supplementation during the ovarian stimulation:

  * were selected for a GnRH agonist protocol to induce pituitary desensitization
  * previous poor ovarian response to r-hFSH alone
  * aged 35 to 40 years
  * elevated baseline hormone parameters that were predictive of poor ovarian response
* Female subjects aged between 18-40 years
* Subjects with uterine cavity able to sustain embryo implantation or pregnancy
* Subject who had no known infection with human immunodeficiency virus, hepatitis B or C virus
* Subjects who were willing to participate and comply with the protocol for the duration of the study
* Subjects who had given informed consent, prior to any study-related procedure not part of normal medical care

Exclusion Criteria:

* Subjects with clinically significant systemic disease (e.g. insulin-dependent diabetes, epilepsy, severe migraine, intermittent porphyria, hepatic, renal or cardiovascular disease, severe corticosteroid-dependent asthma)
* Any contraindication to being pregnant and/or carrying a pregnancy to term
* Subjects with abnormal gynecological bleeding of undetermined origin
* Subjects with known allergy to gonadotrophin preparations
* Subjects with any medical condition for which the use of gonadotrophin preparations was contraindicated
* Subjects who had previously entered into this study or simultaneously participated in another clinical drug trial
* Subjects with any active substance abuse or history of drug, medication or alcohol abuse in the past 5 years
* Subjects who had refused or were unable to comply with protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2004-09; Primary Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Canada Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 4 study centers in Canada from September 2004 to October 2005.
Pre-assignment Details: 55 participants were enrolled in the study, 3 participants discontinued prior to study drug administration as they did not meet the eligibility criteria.
Groups:
- Recombinant Human-Luteinizing Hormone (Luveris): All participants received Luveris 150 International Unit (IU) per day, subcutaneously (s.c) from stimulation day 6 (Day S6) of their assisted reproductive technology (ART) treatment cycle, continuing at the same dose until injection of hCG upto and including day of last FSH dose.
Period: Overall Study
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Started | 52 (Number of participants treated)
Completed | 46
Not Completed | 6
Not completed — Lack of Ovarian Response | 2
Not completed — No Oocytes Retrieved | 3
Not completed — No Fertilization | 1

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 52
Age Continuous [Mean (Standard Deviation); unit: years] | 34.6 (3.6)
Age, Customized [Number; unit: participants]
  <35 years | 22
  >=35 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3
  White | 47
  Hispanic | 1
  Aboriginal | 1
Region of Enrollment [Number; unit: participants]
  Canada | 52
Smoking [Number; unit: participants] — Consumption of cigarettes is inclusive of cigarillos and cigars.
  participants
    0 cigarettes per day | 50
    6-20 cigarettes per day | 1
    >20 cigarettes per day | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Metaphase II Oocytes Per Participant Who Underwent Ovum Pick up for Intra-cytoplasmic Sperm Injection (ICSI)
Description: Mean number of metaphase II oocytes was calculated for each participant undergoing ovum pick up for ICSI. ICSI is an in-vitro fertilization procedure in which a single sperm is injected directly into an egg under a microscope. Metaphase II stage of the oocyte was classified as the time at which the first polar body was observed microscopically. Metaphase II oocytes are a sub-group of the total number of oocytes.
Time Frame: On the day of ovum pick up (Day 1 or 2 after human chorionic gonadotropin [hCG] administration).
Population: Analysis population includes those participants undergoing ICSI whose oocytes were assessed for maturity (Metaphase II) using a microscope.
Measure: Mean (Standard Deviation); unit: Metaphase II Oocytes
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 22
Metaphase II Oocytes | 9.5 (4.2)

2. Primary Outcome: Mean Number of Mature Oocytes Per Participant Who Underwent Ovum Pick up for In Vitro Fertilization (IVF)
Description: Mean number of oocytes undergoing ovum pick up for IVF were calculated for each participant. IVF is a process by which egg cells are fertilized by sperm outside the body, in-vitro.
Time Frame: On the day of ovum pick up (Day 1 or 2 after hCG administration).
Population: Analysis population includes those participants undergoing IVF whose oocytes were assessed for maturity. Mature oocytes can be considered as Metaphase II oocytes.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 4
oocytes | 7.5 (6.8)

3. Secondary Outcome: Mean Number of Oocytes Retrieved Per Number of Follicles Aspirated on the Day of Ovum Pick up
Description: Mean number of oocytes retrieved per number of follicles aspirated on the day of ovum pick up was calculated. Oocyte retrieval is a technique used in in vitro fertilization in order to remove oocytes from the ovary of the female, enabling fertilization outside the body.
Time Frame: On day of ovum pick up (Day 1 or 2 after hCG administration)
Population: ITT population: all participants who received at least one dose of the study drug and underwent vaginal ovum pick up.
Measure: Mean (Standard Deviation); unit: oocytes per aspirated follicle
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 50
oocytes per aspirated follicle | 0.9 (0.2)

4. Secondary Outcome: Number of Participants With Confirmed Pregnancies: Biochemical Pregnancies and Clinical Pregnancies
Description: Biochemical pregnancy: A positive pregnancy test defined as hCG level >10 IU/L in a sample taken at least 14 days after Day 3 embryo transfer or 12 days after Day 5/6 embryo transfer with no further ultrasound confirmation of the existence of a gestational sac in the uterus. Clinical pregnancy: Existence of at least one ultrasonography confirmed gestational sac in the uterus, with or without heartbeat.
Time Frame: Post-hCG days 15-20 and post-hCG days 35-42.
Population: ITT population: all participants who received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 52
participants
  Participants with confirmed biochemical pregnancy | 22
  Participants with confirmed clinical pregnancy | 14

5. Secondary Outcome: Number of Participants With Multiple Pregnancies
Description: Multiple pregnancy is a pregnancy where more than one fetus develops simultaneously in the womb. There are two types of twinning-identical and fraternal. Identical twins represent the splitting of a single fertilized zygote (union of two gametes or male/female sex cells that produce a developing fetus) into two separate individuals.
Time Frame: Post-hCG Day 35-42.
Population: ITT population: all participants who received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 52
participants | 4

6. Secondary Outcome: Number of Live Births
Description: A live birth occurs when a fetus, whatever its gestational age, exits the maternal body and subsequently shows any sign of life, such as voluntary movement, heartbeat, or pulsation of the umbilical cord, for however brief a time and regardless of whether the umbilical cord or placenta are intact.
Time Frame: Post-hCG days 15-20 to pregnancy follow up.
Population: ITT population: all participants who received at least one dose of the study drug.
Measure: Number; unit: Live births
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 52
Live births | 13

7. Secondary Outcome: Pregnancy Loss Per Clinical Pregnancy
Description: Preclinical miscarriage: Spontaneous cessation of a biochemical pregnancy. Early spontaneous abortion: Any spontaneous abortion occurring after confirmation of clinical pregnancy and before completion of 12 weeks of gestation. Late spontaneous abortion: any spontaneous abortion occurring between completion of 12 weeks of gestation and prior to a viable stage. Pregnancy loss per clinical pregnancy was measured as a percentage.
Time Frame: Post-hCG days 35-42.
Population: Participants with confirmed clinical pregnancies.
Measure: Number; unit: Percentage of pregnancy loss
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 14
Percentage of pregnancy loss | 7.14

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Study Drug Discontinuation.
Description: AEs: Any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. TEAEs: AEs that occur during treatment with the study drug. It also included incidences of mild, moderate and severe ovarian hyperstimulation syndrome (OHSS). SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued from the study due to AE were also recorded.
Time Frame: From stimulation Day 1 (S1) to post-hCG days 35-42 (safety visit).
Population: ITT population: all participants who received at least one dose of the study drug.
Measure: Number; unit: Number of participants
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 52
Number of participants
  TEAEs | 15
  SAEs | 3
  Discontinuation due to AEs | 0

ADVERSE EVENTS:
Time Frame: AEs are collected on an ongoing basis from day of written informed consent. All new AEs must be recorded until the post-treatment safety, on day 35-42 post-hCG administration. AEs are classified as pre-treatment, treatment-emergent and post-treatment.
Description: Pre-Treatment:Medical conditions present at the initial study visit that did not worsen in severity or frequency during the study;Treatment-Emergent: If the onset date of the AE was on or after the first dose date of the study medication; Post-Treatment: If the onset date of the AE was post-hCG Days 15- 42 for participants who completed the study.
Arm/Group | Recombinant Human-Luteinizing Hormone (Luveris)
Serious Adverse Events (participants affected / at risk) | 3/52
Other Adverse Events (participants affected / at risk) | 15/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recombinant Human-Luteinizing Hormone (Luveris) (N=52)
Abdominal pain (Gastrointestinal disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recombinant Human-Luteinizing Hormone (Luveris) (N=52)
Local tolerability of injections (General disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Injection site pain (General disorders) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Post procedural nausea (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Procedural vomiting (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1
Anxiety (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Genital pruritus female (Reproductive system and breast disorders) | 1
Ovarian Hyperstimulation Syndrome (Reproductive system and breast disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other